CLINICAL TRIAL: NCT04930705
Title: Prospective Clinical Study To Assess The Safety And Efficacy Of The Tempsure Flexsure Applicators For The Treatment Of Abdominal Wrinkles
Brief Title: Study To Assess The Safety And Efficacy Of The Tempsure Flexsure Applicators For Abdominal Wrinkles
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: This study was terminated because of a business decision.
Sponsor: Cynosure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7027-PL01-2021
Record Dates: First submitted 2021-06-11; First posted 2021-06-18 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Wrinkle
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- TempSure FlexSure Applicator (Experimental): Subjects will be treated with the TempSure FlexSure applicator device at each treatment.
  Interventions: Device: Treatment with TempSure Applicator

INTERVENTIONS:
Device: Treatment with TempSure Applicator — Subjects will receive up to 5 treatments on the abdomen.

SUMMARY:
Subjects will be enrolled at 1 study center. Subjects may receive 5 treatments with the TempSure® device on the abdomen for wrinkles.

ELIGIBILITY:
Inclusion Criteria:

* A healthy, non-smoking male or female between the age of 18 - 55 years old.
* Willing to receive treatments with the TempSure® device.
* Understand and accept obligation not to receive any other procedures on the treatment and control area throughout the length of the study.
* Understands and accepts the obligation and is logistically able to be present for all visits.
* Is willing to comply with all requirements of the study and sign the informed consent document.

Exclusion Criteria:

* Is pregnant or of child bearing potential and not using medically effective birth control, or has been pregnant in the last 3 months, currently breast feeding or planning a pregnancy during the study.
* The subject is currently enrolled in an investigational drug or device trial or has received an investigational drug or been treated with an investigational device within in the area to be treated 6 months prior to entering this study.
* The subject has a cut, wound, or infected skin on the area to be treated.
* The subject is on local, oral, or systemic anesthetic agents.
* The subject has nerve insensitivity to heat in the treatment area.
* The subject has any condition or is in a situation which in the investigators opinion may put the subject at significant risk, may confound study results or may interfere significantly with the subject's participation.

Cautionary Criteria:

* The subject has any embedded electronic device that gives or receives a signal, the device should be turned off or removed prior to treatment.
* The subject has an embedded pacemaker or implantable cardioverter defibrillator (ICD), the client's cardiologist must be consulted prior to treatment.

NOTE: This device has not been tested on patients implanted with electronic devices that receive or emit signals, such as: Pacemakers, Implantable Cardiac Defibrillators (ICD), or Cardiac Resynchronization Therapy (CRT) devices.

* If the neutral pad would need to be placed on a subject that has a metal plate, rod, or any metal implant that could conduct heat from the Smart Handpiece or surgical handpiece.
* The subject is allergic to adhesives, such as glues on medical tape, they should be alerted that a rash may occur on the neutral pad site and an over the counter solution may be used to treat the area.
* If the subject has an unhealthy expectation of the results - this is not plastic surgery and all subject should be fully informed of the treatment's expected results.
* The subject has severe laxity or sagging that causes redundant folds of tissue or hanging skin in the area to be treated - this treatment will be ineffective.
* The subject has used Accutane (Isotretinoin) six to twelve months prior to treatment, as this can thin the skin and make it britlle
* Studies of the use of the RF generator on subjects that have any of the following conditions is unknown:

  * Autoimmune Disease
  * Diabetic
  * Herpes Simplex
* Use caution when treating areas that have tattoos, permanent makeup, and permanent brows.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Correct Identification of Pre-Treatment Images Compared to Follow Up Images | 30 Day Follow Up
  Blinded independent reviewers will be given pre-treatment and 30 day follow up images and will identify which image is pre-treatment, and which image was taken at the follow up. The percentage of correct images identified will be reported.
Correct Identification of Pre-Treatment Images Compared to Follow Up Images | 90 Day Follow Up
  Blinded independent reviewers will be given pre-treatment and 90 day follow up images and will identify which image is pre-treatment, and which image was taken at the follow up. The percentage of correct images identified will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Civiok, Study Director — Cynosure, Inc.
Locations (1):
- JUVA Skin & Laser Center, New York, New York, United States